CLINICAL TRIAL: NCT04464980
Title: NIDA-CTN-0100: Optimizing Retention, Duration and Discontinuation Strategies for Opioid Use Disorder Pharmacotherapy (RDD)
Brief Title: Optimizing Retention, Duration and Discontinuation Strategies for Opioid Use Disorder Pharmacotherapy (RDD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York State Psychiatric Institute (Other); Columbia University (Other); Harvard Medical School (HMS and HSDM) (Other); Mclean Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 19-01363; CTN-0100 (Other: NIDA Clinical Trials Network); UG1DA013035 (NIH); UG1DA015831 (NIH); 20-PRS-057 (Other: Biomedical Research Alliance of New York (BRANY) sIRB); 146193 (Other: FDA/IND#)
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder (OUD)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine; vivitrol

STUDY DESIGN:
Intervention Model Description: Retention Phase: 3x2 for BUP; 1x2 for XR-NTX; Discontinuation Phase: 2x2 for SL-BUP; 1x2 for XR-BUP; 1x2 for XR-NTX
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Retention: SL-BUP standard dose + MM (Experimental): Standard dose sublingual buprenorphine-naloxone (SL-BUP) 16mg/day target plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: SL-BUP; Behavioral: MM
- Retention: SL-BUP high dose + MM (Experimental): High dose sublingual buprenorphine-naloxone (SL-BUP) 32mg/day target plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: SL-BUP; Behavioral: MM
- Retention: XR-BUP + MM (Experimental): Extended-release injectable buprenorphine (XR-BUP) plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: XR-BUP; Behavioral: MM
- Retention: XR-NTX + MM (Experimental): Extended-release injectable naltrexone (XR-NTX) plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: XR-NTX; Behavioral: MM
- Retention: SL-BUP standard dose + MMR (Experimental): Standard dose sublingual buprenorphine-naloxone (SL-BUP) 16mg/day target plus MMR, consisting of Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: SL-BUP; Behavioral: MMR
- Retention: SL-BUP high dose + MMR (Experimental): High dose sublingual buprenorphine-naloxone (SL-BUP) 32mg/day target plus MMR, consisting of standard Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: SL-BUP; Behavioral: MMR
- Retention: XR-BUP + MMR (Experimental): Extended-release injectable buprenorphine (XR-BUP) plus MMR, consisting of standard Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: XR-BUP; Behavioral: MMR
- Retention: XR-NTX + MMR (Experimental): Extended-release injectable naltrexone (XR-NTX) plus MMR, consisting of standard Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: XR-NTX; Behavioral: MMR
- Discontinuation: Discontinue SL-BUP with SL-BUP + MM (Experimental): Start on SL-BUP, taper with SL-BUP, plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: SL-BUP; Behavioral: MM
- Discontinuation: Discontinue SL-BUP with XR-BUP + MM (Experimental): Start on SL-BUP, taper with XR-BUP, plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: XR-BUP; Behavioral: MM
- Discontinuation: Discontinue XR-BUP with XR-BUP + MM (Experimental): Start on XR-BUP, taper with XR-BUP, plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: XR-BUP; Behavioral: MM
- Discontinuation: Discontinue XR-NTX with XR-NTX + MM (Experimental): Start on XR-NTX, taper with XR-NTX, plus MM, consisting of standard Medical Management and usual counseling at the treatment program.
  Interventions: Drug: XR-NTX; Behavioral: MM
- Discontinuation: Discontinue SL-BUP with SL-BUP + MMD (Experimental): Start on SL-BUP, taper with SL-BUP, plus MMD, consisting of standard Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: SL-BUP; Behavioral: MMD
- Discontinuation: Discontinue SL-BUP with XR-BUP + MMD (Experimental): Start on SL-BUP, taper with XR-BUP, plus MMD, consisting of standard Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: XR-BUP; Behavioral: MMD
- Discontinuation: Discontinue XR-BUP with XR-BUP + MMD (Experimental): Start on XR-BUP, taper with XR-BUP, plus MMD, consisting of standard Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: XR-BUP; Behavioral: MMD
- Discontinuation: Discontinue XR-NTX with XR-NTX + MMD (Experimental): Start on XR-NTX, taper with XR-NTX, plus MMD, consisting of standard Medical Management and usual counseling, plus a technology-based behavioral component.
  Interventions: Drug: XR-NTX; Behavioral: MMD

INTERVENTIONS:
Drug: SL-BUP — Daily dosing of sublingual buprenorphine-naloxone
  Other Names: sublingual buprenorphine; Suboxone
  Arms: Discontinuation: Discontinue SL-BUP with SL-BUP + MM; Discontinuation: Discontinue SL-BUP with SL-BUP + MMD; Retention: SL-BUP high dose + MM; Retention: SL-BUP high dose + MMR; Retention: SL-BUP standard dose + MM; Retention: SL-BUP standard dose + MMR
Drug: XR-BUP — Weekly/monthly dosing of extended-release injectable buprenorphine
  Other Names: extended-release buprenorphine; CAM2038; Brixadi
  Arms: Discontinuation: Discontinue SL-BUP with XR-BUP + MM; Discontinuation: Discontinue SL-BUP with XR-BUP + MMD; Discontinuation: Discontinue XR-BUP with XR-BUP + MM; Discontinuation: Discontinue XR-BUP with XR-BUP + MMD; Retention: XR-BUP + MM; Retention: XR-BUP + MMR
Drug: XR-NTX — Monthly dosing of extended-release injectable naltrexone
  Other Names: extended-release naltrexone; Vivitrol
  Arms: Discontinuation: Discontinue XR-NTX with XR-NTX + MM; Discontinuation: Discontinue XR-NTX with XR-NTX + MMD; Retention: XR-NTX + MM; Retention: XR-NTX + MMR
Behavioral: MM — MM consists of standard Medical Management and the usual counseling at the treatment program.
  Arms: Discontinuation: Discontinue SL-BUP with SL-BUP + MM; Discontinuation: Discontinue SL-BUP with XR-BUP + MM; Discontinuation: Discontinue XR-BUP with XR-BUP + MM; Discontinuation: Discontinue XR-NTX with XR-NTX + MM; Retention: SL-BUP high dose + MM; Retention: SL-BUP standard dose + MM; Retention: XR-BUP + MM; Retention: XR-NTX + MM
Behavioral: MMR — MMR consists of Medical Management and usual counseling, plus a technology-based behavioral component.
  Arms: Retention: SL-BUP high dose + MMR; Retention: SL-BUP standard dose + MMR; Retention: XR-BUP + MMR; Retention: XR-NTX + MMR
Behavioral: MMD — MMD consists of Medical Management and usual counseling, plus a technology-based behavioral component.
  Arms: Discontinuation: Discontinue SL-BUP with SL-BUP + MMD; Discontinuation: Discontinue SL-BUP with XR-BUP + MMD; Discontinuation: Discontinue XR-BUP with XR-BUP + MMD; Discontinuation: Discontinue XR-NTX with XR-NTX + MMD

SUMMARY:
This is a two phase study investigating combinations of pharmacological and behavioral interventions to optimize the treatment of Opioid Use Disorder (OUD). The Retention Phase will assess strategies for improving retention on buprenorphine (BUP) and extended-release injectable naltrexone (XR-NTX). The Discontinuation Phase will assess which approaches are most likely to lead to long-term success (absence of relapse), and what characteristics of participants distinguish those who can safely discontinue Medications for Opioid Use Disorder (MOUD) from those who remain at risk of relapse and should not discontinue.

DETAILED DESCRIPTION:
The main objectives of this study are:

1. To test strategies to improve retention in treatment on medications for opioid use disorder (MOUD), among patients initiating treatment for OUD.
2. To test strategies to improve outcomes among patients who have achieved stable remission on MOUD and want to discontinue MOUD.
3. To develop models to predict who is able to discontinue MOUD without relapse, based on patient characteristics, including duration of MOUD prior to discontinuation.

The study will have a multicenter, randomized, pragmatic non-blinded design. The study has two phases, a Retention Phase and a Discontinuation Phase.

ELIGIBILITY:
Inclusion Criteria for Retention Phase:

1. 18 years of age or older;
2. Meet DSM-5 criteria for current opioid use disorder (heroin, fentanyl or other synthetic opioids, and/or prescription opioids);
3. Seeking treatment for opioid use disorder and choosing either buprenorphine (BUP) or extended-release injection naltrexone (XR-NTX);
4. If choosing buprenorphine, willing to be randomized to SL-BUP-16mg, SL-BUP-32mg, or XR-BUP;
5. Willing to be randomized to either MM (standard Medical Management plus counseling treatment as usual available at the site) or MMR (MM plus usual counseling and access to an app delivering CM + CBT);
6. In good-enough general health (meaning good enough health to be in outpatient treatment) as determined by the study medical clinician on the basis of medical history, review of systems, and physical/mental status exam, to permit treatment with XR-NTX or BUP;
7. Willing and able to provide written informed consent;
8. Able to speak English sufficiently to understand the study procedures;
9. If female of childbearing potential, willing to practice an effective method of birth control for the duration of participation in the study (participants who become pregnant during the study will continue to be followed; treatment may be modified consistent with pregnancy).

Exclusion Criteria for Retention Phase:

1. Serious medical, psychiatric, or co-occurring substance use disorder or concomitant medication that, in the opinion of the study medical clinician, makes the patient not appropriate for outpatient treatment with buprenorphine or XR-NTX, but instead requires a higher or different level of care. Examples include:

   1. Disabling or terminal medical illness (e.g., uncompensated heart failure, cirrhosis or end-stage liver disease) as assessed by medical history, review of systems, physical exam and/or laboratory assessments;
   2. Severe, untreated or inadequately treated psychiatric condition (e.g., active psychosis, uncontrolled bipolar disorder) as assessed by history and/or clinical interview, requiring a different level of care (e.g., hospitalization);
   3. Current severe alcohol, benzodiazepine, or other depressant or sedative hypnotic use, requiring a different level of care (e.g., hospitalization);
2. Suicidal or homicidal ideation or behavior requiring a different level of care (e.g., hospitalization);
3. Known allergy or sensitivity to preferred medication or its components;
4. Maintenance on methadone at the time of signing consent;
5. For those preferring XR-NTX, presence of pain of sufficient severity as to require ongoing pain management with opioids;
6. For those preferring XR-NTX, body habitus that, in the judgment of the study physician, precludes safe intramuscular injection of XR-NTX (e.g., BMI>40, excess fat tissue over the buttocks, emaciation);
7. If female, currently pregnant or breastfeeding or planning on conception;
8. Are currently in jail, prison or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities;
9. Have used the reSET-O or CHESS Connections mHealth apps in the 3 months prior to consent;
10. Other major reasons that might prevent an individual from participating in the study (e.g., a planned move out of the area).

Inclusion Criteria for Discontinuation Phase:

1. 18 years of age or older;
2. Have been receiving buprenorphine for OUD for at least the past year or XR-NTX pharmacotherapy for OUD for at least the past 6 months prior to consent for the Discontinuation Phase;
3. Express the desire to discontinue MOUD after a shared decision-making discussion with the treating provider;
4. Meet stability criteria, i.e., have abstained from opioids (other than buprenorphine), cocaine, methamphetamine, and non-prescribed benzodiazepines for the past ≥12 weeks, and do not meet DSM-5 criteria for current (≥12 weeks) alcohol use disorder (participants with cannabis use will be eligible);
5. If currently taking buprenorphine, are willing to take either SL-BUP or XR-BUP if randomized to that condition;
6. Willing to be randomized to either MM or to MMD;
7. Able to provide written informed consent after discussion with their provider regarding the risks of discontinuation;
8. Able to speak English sufficiently to understand the study procedures;
9. If female of childbearing potential, willing to practice an effective method of birth control while in the study and taking study medication (participants who become pregnant during the study will continue to be followed; treatment may be modified consistent with pregnancy).

Exclusion Criteria for Discontinuation Phase:

1. Serious medical or psychiatric disorder or concomitant medication that, in the opinion of the study medical clinician, would make study participation hazardous to the participant or compromise study findings or would prevent the participant from completing the study. Examples include:

   1. Disabling or terminal medical illness (e.g., uncompensated heart failure, cirrhosis or end-stage liver disease) as assessed by medical history, review of systems, physical exam and/or laboratory assessments;
   2. Severe, untreated, or inadequately treated psychiatric condition (e.g., active psychosis, uncontrolled bipolar disorder) as assessed by history and/or clinical interview, requiring a different level of care (e.g., hospitalization);
2. Suicidal or homicidal ideation or behavior requiring a different level of care (e.g., hospitalization);
3. For participants entering the study taking buprenorphine, presence of pain requiring or likely requiring ongoing pain management with buprenorphine or other opioids;
4. If female, currently pregnant or breastfeeding or planning on conception;
5. Use of opioids (other than buprenorphine), cocaine, methamphetamine, or non-prescribed benzodiazepines in the past 12 weeks;
6. Meets current DSM-5 criteria for any current alcohol use disorder;
7. Are currently in jail, prison or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities;
8. Have used the Connections mHealth app in the 3 months prior to consent (other than Connections in the Retention Phase);
9. Other major reasons that might prevent an individual from participating in the study (e.g., a planned move out of the area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Retention: Continuous retention in MOUD treatment at 26 weeks | Retention: at week 26
  Binary (yes/no). Continuously enrolled in maintenance treatment on one or more of the evidence-based MOUD modalities (e.g., SL-BUP, XR-BUP, XR-NTX, or methadone maintenance) with no more than a 28-day gap in MOUD over the 26-week period.
Discontinuation: Completed Discontinuation without Relapse | Discontinuation: at week 24 follow up
  Binary (yes/no). Discontinuing MOUD during the taper period, no return to MOUD, and no relapse to opioid use, either during the taper (up to 48 weeks for those entering on BUP or 24 weeks for those entering on XR-NTX) or during the 24 weeks after MOUD is discontinued.

SECONDARY OUTCOMES:
Retention KS1: Weekly opioid abstinence | Retention: through week 26
  Weekly opioid abstinence (measured by Timeline Followback, not contradicted by toxicology test). Repeated yes/no measure for each of weeks 3 through 26.
Retention KS2: Treatment effectiveness | Retention: at week 26
  Retention treatment effectiveness, measured by the Treatment Effectiveness Assessment (TEA, Ling et. al, 2012); a brief instrument to assess patient progress in treatment and recovery along 4 domains (substance use, health, lifestyle and community) at week 26.
Discontinuation KS1: Other discontinuation outcomes | Discontinuation: at week 24 follow up
  Participants who did not meet the criteria for the primary outcome (Completed Discontinuation without Relapse), will be subcategorized into 3 other outcome categories: 1) Did not Complete Discontinuation (i.e., MOUD is continued or discontinued and then restarted within the next 24 weeks) and did not Relapse; 2) Completed Discontinuation followed by Relapse; or 3) Did not Complete Discontinuation and Relapse (i.e., relapse while on MOUD).
DSK2: Treatment effectiveness | Discontinuation: week 24 follow up
  Discontinuation treatment effectiveness, measured by the Treatment Effectiveness Assessment (TEA, Ling et. al, 2012); a brief instrument to assess patient progress in treatment and recovery along 4 domains (substance use, health, lifestyle and community) at week 24. Measured at the end of taper (EOT): up to 24 weeks for tapers with XR-NTX and up to 48 weeks for tapers with BUP; and at the week 24 follow up (primary outcome timepoint).

OTHER OUTCOMES:
R-Other 1a: Continuous opioid abstinence-weeks 23-26 | Retention: weeks 23-26
  Binary indicator of continuous abstinence from opioids in weeks 23 to 26 (measured by Timeline Followback, not contradicted by toxicology test)
R-Other 1b: Continuous opioid abstinence-weeks 47-50 | Retention: weeks 47-50
  Binary indicator of continuous abstinence from opioids in weeks 47 to 50 (measured by Timeline Followback, not contradicted by toxicology test)
R-Other 1c: Continuous opioid abstinence-weeks 71-74 | Retention: weeks 71-74
  Binary indicator of continuous abstinence from opioids in weeks 71 to 74 (measured by Timeline Followback, not contradicted by toxicology test)
R-Other 2: Weekly opioid abstinence | Retention: weeks 27-74
  Weekly opioid abstinence (measured by Timeline Followback, not contradicted by toxicology test). Repeated yes/no measure for each of weeks 27 through 74.
R-Other 3: Weekly abstinence from other substance use | Retention: weeks 0-74
  Weekly abstinence from other substance use (measured by Timeline Followback, not contradicted by toxicology test)
R-Other 4: Craving | Retention: weeks 0-98
  Craving, measured by the Opioid Craving Scale
R-Other 5a: Stable abstinence at week 26 | Retention: week 26
  Stable abstinence, as defined by the same stability criteria as in the Discontinuation Phase (point prevalence stability at week 26), i.e., past ≥12 weeks of consecutive abstinence from opioids (other than prescribed buprenorphine), methamphetamine, and cocaine, no non-prescribed benzodiazepine use, and no current (≥12 weeks) alcohol use disorder (any severity); measured by Timeline Followback, not contradicted by toxicology test (both repeated measures), and DSM-5 checklist for current alcohol use disorder (which is performed only when these abstinence criteria are met)
R-Other 5b: Stable abstinence at week 50 | Retention: week 50
  Stable abstinence, as defined by the same stability criteria as in the Discontinuation Phase (point prevalence stability at week 50), i.e., past ≥12 weeks of consecutive abstinence from opioids (other than prescribed buprenorphine), methamphetamine, and cocaine, no non-prescribed benzodiazepine use, and no current (≥12 weeks) alcohol use disorder (any severity); measured by Timeline Followback, not contradicted by toxicology test (both repeated measures), and DSM-5 checklist for current alcohol use disorder (which is performed only when these abstinence criteria are met)
R-Other 5c: Stable abstinence at week 74 | Retention: week 74
  Stable abstinence, as defined by the same stability criteria as in the Discontinuation Phase (point prevalence stability at week 74), i.e., past ≥12 weeks of consecutive abstinence from opioids (other than prescribed buprenorphine), methamphetamine, and cocaine, no non-prescribed benzodiazepine use, and no current (≥12 weeks) alcohol use disorder (any severity); measured by Timeline Followback, not contradicted by toxicology test (both repeated measures), and DSM-5 checklist for current alcohol use disorder (which is performed only when these abstinence criteria are met)
R-Other 6: Retention in MOUD at week 50 | Retention: week 50
  Point prevalence of retention in MOUD treatment (defined as no gap of 28 days or more in MOUD) at 50 weeks after date of randomization (binary, measured by Timeline Followback)
R-Other 7: Retention in MOUD at week 74 | Retention: week 74
  Point prevalence of retention in MOUD treatment at 74 weeks after date of randomization, measured by TLFB
R-Other 8: Dropout from MOUD treatment | Retention: weeks 0-74
  Dropout from MOUD treatment (time to event), i.e., a gap of 28 or more days in MOUD, event to have started at the beginning of the 28-day gap (measured by Timeline Followback)
R-Other 9: Depression | Retention: weeks 0-26
  Depression (measured by the Patient Health Questionnaire (PHQ) 9) over the first 26 weeks
R-Other 10: Anxiety | Retention: weeks 0-26
  Anxiety, measured by the measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Preference (PROPr) over the first 26 weeks
R-Other 11: Stress | Retention: weeks 0-26
  Stress, measured by the Perceived Stress Scale, over the first 26 weeks
R-Other 12: Pain | Retention: weeks 0-26
  Pain, measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Preference (PROPr), over the first 26 weeks
R-Other 13: Recovery capital | Retention: weeks 0-26
  Recovery capital, measured by the Brief Assessment of Recovery Capital (BARC) 10 item scale, over the first 26 weeks
R-Other 14: Negative consequences of opioid use | Retention: weeks 0-26
  Negative consequences of opioid use, measured by the Short Inventory of Problems-Revised, over the first 26 weeks
R-Other 15: Sexual risk | Retention: weeks 0-26
  Sexual risk, measured by two questions regarding sexual behavior, over the first 26 weeks
R-Other 16: Rate of incarceration | Retention: weeks 0-26
  Rate of incarcerations, collected on the Non-Medical and Other Services form, over the first 26 weeks
R-Other 17: Rate of homelessness | Retention: weeks 0-26
  Rate of homelessness, collected on the Study Demographics form, over the first 26 weeks
D-Other 1: Relapse | Discontinuation: during taper and through week 24 follow up
  Relapse (time to event): defined as self-reported opioid use on more than 4 days in any consecutive 28-day period (event to begin on the first day of use), or 2 or more consecutive opioid-positive drug tests (event to begin with the first opioid-positive test) or any self-reported injection drug use (whichever comes first).
D-Other 2: Withdrawal symptoms | Discontinuation: during taper and through week 24 follow up
  Withdrawal symptoms, measured by Subjective Opioid Withdrawal Scale (SOWS), during taper and follow up
D-Other 3: Craving | Discontinuation: during taper and through week 24 follow up
  Craving, measured by the Opioid Craving Scale, during taper and follow up
D-Other 4: Depression | Discontinuation: during taper and through week 24 follow up
  Depression, measured by the Patient Health Questionnaire (PHQ) 9 item, during taper and follow up
D-Other 5: Anxiety | Discontinuation: during taper and through week 24 follow up
  Anxiety, measured by the measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Preference (PROPr), during taper and follow up
D-Other 6: Stress | Discontinuation: during taper and through week 24 follow up
  Stress, measured by the Perceived Stress Scale, during taper and follow up
D-Other 7: Pain | Discontinuation: during taper and through week 24 follow up
  Pain, measured by the measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Preference (PROPr), during taper and follow up
D-Other 8a: Recovery capital (BARC-10) | Discontinuation: during taper and through week 24 follow up
  Recovery capital, measured by the Brief Assessment of Recovery Capital (BARC) 10 item scale, during taper and follow up
D-Other 8b: Recovery capital (RCS) | Discontinuation: during taper and through week 24 follow up
  Recovery capital, measured by the Recovery Capital Scale; six additional questions more specific to participants with OUD, during taper and follow up
D-Other 9: Negative consequences of opioid use | Discontinuation: during taper and through week 24 follow up
  Negative consequences of opioid use, measured by the Short Inventory of Problems-Revised, during taper and follow up
D-Other 10: Sexual risk | Discontinuation: during taper and through week 24 follow up
  Sexual risk, measured by two questions regarding sexual behavior, during taper and follow up
D-Other 11: Rate of incarceration | Discontinuation: during taper and through week 24 follow up
  Incarcerations, collected on the Non-Medical and Other Services form, during taper and follow up
D-Other 12: Rate of homelessness | Discontinuation: during taper and through week 24 follow up
  Homelessness, collected on the Study Demographics form, during taper and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Edward V Nunes, MD, Principal Investigator — New York State Psychiatric Institute/Columbia University Irving Medical Center; John Rotrosen, MD, Principal Investigator — NYU Langone Health; Roger Weiss, MD, Principal Investigator — Harvard Medical School/McLean Hospital
Locations (21):
- United States (21):
  - University of Arkansas for Medical Sciences (UAMS) / Center for Addiction Services and Treatment (CAST), Little Rock, Arkansas
  - Tarzana Treatment Centers, Inc., Tarzana, California
  - Liberation Programs, Inc., Bridgeport, Connecticut
  - Operation PAR, Clearwater, Florida
  - Gateway Community Services, Jacksonville, Florida
  - Aspire Health Partners, Orlando, Florida
  - Mountain Manor / Maryland Treatment Centers, Baltimore, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Stanley Street Treatment and Resources, Inc., Fall River, Massachusetts
  - Square Medical Group, LLC, Newton, Massachusetts
  - Gibson Center for Behavioral Change, Cape Girardeau, Missouri
  - Dartmouth Hitchcock - ATP, Lebanon, New Hampshire
  - University of New Mexico Addiction and Substance Abuse Program, Albuquerque, New Mexico
  - Bellevue Hospital Center, New York, New York
  - Adapt Integrated Health Care, Roseburg, Oregon
  - Adapt Integrated Health Care, Winston, Oregon
  - Center for Psychiatric and Chemical Dependency Services (CPCDS), Pittsburgh, Pennsylvania
  - Internal Medicine Recovery Engagement Program (IM-REP), Pittsburgh, Pennsylvania
  - Shoreline Behavioral Health Services, Conway, South Carolina
  - Huntsman Mental Health Institute / University of Utah, Salt Lake City, Utah
  - Chestnut Ridge Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Implementation Guidance (https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm) and (for HEAL-funded studies) the HEAL Public Access and Data Sharing Policy (https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/research/heal-public-access-data-sharing-policy).
  Primary data for this study will be available to the public in the NIDA data repository. For more details on data sharing please visit https://datashare.nida.nih.gov/.
  The primary outcome(s) publication will be included along with study underlying primary data in the data share repository, and it will also be deposited in PubMed Central http://www.pubmedcentral.nih.gov/ per NIH Policy (http://publicaccess.nih.gov/).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
URL: https://datashare.nida.nih.gov

REFERENCES:
- [Derived] Shulman M, Meyers-Ohki S, Novo P, Provost S, Ohrtman K, Van Veldhuisen P, Oden N, Otterstatter M, Bailey GL, Liu D, Rotrosen J, Weiss RD, Nunes EV. Optimizing retention strategies for opioid use disorder pharmacotherapy: The retention phase of the CTN-0100 trial (RDD). Contemp Clin Trials. 2025 Mar;150:107816. doi: 10.1016/j.cct.2025.107816. Epub 2025 Jan 20. PMID 39842691
- [Derived] Shulman M, Provost S, Ohrtman K, Novo P, Meyers-Ohki S, Van Veldhuisen P, Oden N, Otterstatter M, Bailey GL, Liu D, Rotrosen J, Nunes EV, Weiss RD. Discontinuation of medication treatment for opioid use disorder after a successful course: The discontinuation phase of the CTN-0100 (RDD) trial. Contemp Clin Trials. 2024 Jul;142:107543. doi: 10.1016/j.cct.2024.107543. Epub 2024 Apr 23. PMID 38657730

DOCUMENTS (1):
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04464980/ICF_000.pdf